CLINICAL TRIAL: NCT01517269
Title: PETS-D (Parent Education Thru Simulation-Diabetes)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Susan Sullivan-Bolyai, Study Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13643
Record Dates: First submitted 2012-01-13; First posted 2012-01-25 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Type 1 Diabetes
Keywords: Parent education
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education with simulator (Experimental): Parent randomized to this group will be taught diabetes management with vignette and simulator
  Interventions: Behavioral: Parent education with human patient simulator
- Control arm: standard diabetes education (Active Comparator): Parents will receive standard diabetes education with a diabetes educator
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Parent education with human patient simulator — After child is newly diagnosed with Type 1 diabetes, parents will receive 3 teaching sessions over 12 weeks, after baseline data collected, at 1 month, and at 3 months, covering hypoglycemia, hyperglycemia and pattern management using teaching vignettes and practice with human patient simulator
  Arms: Education with simulator
Behavioral: Standard care — After child is newly diagnosed with Type 1 diabetes, parents will receive 3 teaching sessions over 12 weeks, after baseline data collected, at 1 month, and at 3 months, covering hypoglycemia, hyperglycemia and pattern management without the use of a simulator
  Arms: Control arm: standard diabetes education

SUMMARY:
Hypothesis: Parents who receive Parent Education Thru Simulation-Diabetes (PETS-D) will have significantly higher diabetes knowledge (cognitive visual schemata), better technical and problem-solving competence and confidence, and lower fear and stress/anxiety levels; and provide better diabetes management at 14 weeks compared to those parents receiving standard diabetes education.

ELIGIBILITY:
Inclusion Criteria:

* parents 18 years and older who have a child newly diagnosed with type 1 diabetes mellitus (T1DM) from 5 years old to under 13 years of age

Exclusion Criteria:

* exclude children with developmental delays (such as Down Syndrome, Autism) or steroid induced diabetes (cancer treatment related or cystic fibrosis)
* exclude parents who require insulin treatment -or- those that have another child with TIDM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2010-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in baseline of Diabetes Knowledge | Baseline and 14 weeks
  Diabetes Awareness and Reasoning Test-Parents (DART-P)is a 47-item multiple-choice questionnaire. The subscales include general, insulin, hyper-hypglycemia, and problem-solving. Parent education was a significant predictor of total scores.

SECONDARY OUTCOMES:
Change in Baseline of Problem solving | Baseline and 14 weeks
  Wysocki's Modified Problem-solving measure18 (PSM) is a 5 item questionnaire that focuses on how to proactively prevent and treat hypoglycemia. Dr. Wysocki sent us one of his vignettes developed from the structured interview measure. Based on the examples of probes that are part of the interview, we constructed a 5-question multiple choice instrument to measure parental problem-solving abilities and knowledge synthesis. We will report the reliability and validity of this measure with data from the proposed study.
Change in Baseline of Diabetes management | Baseline and 14 weeks
  Diabetes Management Outcomes is a 5 question likert scale based on ADA2 management recommendations.
Change in Baseline of Diabetes self efficacy | Baseline and 14 weeks
  The Self-Efficacy Diabetes-Pediatrics (SED-P) will be used to measure parent confidence in specific task and skill associated diabetes care, i.e. how confident they feel to perform day-to-day diabetes management.
Change in Baseline of Fear of hypoglycemia | Baseline and 14 weeks
  The Hypoglycemia Fear Survey-Parents (HFS-P) total score will be used to measure parental fears and avoidance behaviors associated with hypoglycemia in their children.There are 2 subscales that measure parental concerns of their child experiencing an episode of hypoglycemia and behaviors they use to prevent these episodes from occurring
Change in Baseline of Parent anxiety | Baseline and 14 weeks
  State-Trait Anxiety (STAI) is a well established 40-item instrument (Likert scale, with 1 being not at all, to 4 being almost always) used to measure situational (state, how one feels at this moment) and stable (trait, how one feels in general) tendencies toward anxiety. Higher scores signify more anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts, Worcester, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Sullivan-Bolyai S, Crawford S, Bova C, Lee M, Quintos JB, Johnson K, Cullen K, Hamm T, Bisordi J, Ramchandani N, Fletcher J, Quinn D, Jaffarian C, Lipman T, Melkus G. PETS-D: Impact on Diabetes Management Outcomes. Diabetes Educ. 2015 Oct;41(5):537-49. doi: 10.1177/0145721715598383. Epub 2015 Aug 5. PMID 26246593